CLINICAL TRIAL: NCT00405015
Title: The Effect of Rosiglitazone on Ischemia-reperfusion-injury Using Annexin A5 Scintigraphy. A Double Blind Placebo- Controlled Cross-over Study in Subjects With the Metabolic Syndrome
Brief Title: The Effect of Rosiglitazone on Ischemia-reperfusion-injury Using Annexin A5 Scintigraphy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AR49653-4; EudraCT number 2006-006208-13
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Last update posted 2010-08-24 (Estimated); Status verified 2008-10

CONDITIONS: Ischemia-Reperfusion Injury; The Metabolic Syndrome
Keywords: rosiglitazone; ischemia-reperfusion injury; human; Annexin A5 scintigraphy; metabolic syndrome
MeSH Terms: conditions — Reperfusion Injury; Metabolic Syndrome | interventions — Rosiglitazone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Placebo first
  Interventions: Drug: rosiglitazone
- 2 (Experimental): Rosiglitazone first
  Interventions: Drug: rosiglitazone

INTERVENTIONS:
Drug: rosiglitazone — Rosiglitazone 4 mg bidaily for 8 weeks

SUMMARY:
Cardiovascular disease is the leading cause of death in diabetic patients due to both a high event rate and a worse outcome. A pharmacological intervention that reduces ischemia-reperfusion-injury would improve the outcome of diabetic patients after a cardiovascular event. In the present study, we will use annexinA5 scintigraphy to address the following hypothesis:

Rosiglitazone reduces ischemia-reperfusion-injury in humans with insulin resistance.

DETAILED DESCRIPTION:
Rationale: Cardiovascular disease is the leading cause of death in diabetic patients due to both a high event rate and a worse outcome. A pharmacological intervention that reduces ischemia-reperfusion-injury would improve the outcome of diabetic patients after a cardiovascular event. The thiazolidinedione derivatives are peroxisome proliferator-activated receptor-γ (PPARγ) ligands that are approved for the treatment of hyperglycemia in type 2 diabetes mellitus. Animal data suggest that PPARγ ligands can protect against ischemia-reperfusion-injury by improving insulin responsiveness. However, no human data on these beneficial effects are available. Recently, our group developed a human in vivo model to quantify ischemia-reperfusion-injury. In this model annexin A5 scintigraphy is used to visualize early and reversible cellular membrane changes that occur in the forearm skeletal muscle vascular bed after ischemic exercise. In the present study, we will use this approach to address the following hypothesis: Rosiglitazone reduces ischemia-reperfusion-injury in humans with insulin resistance, selected by using the criteria for the metabolic syndrome.

Study design: This is a single-center randomized, double blind, placebo-controlled crossover study with a washout period of 6 weeks.

Study population: Men and postmenopausal women, age 20-70 years with the metabolic syndrome.

Intervention: Every subject uses during 8 weeks rosiglitazone 4 mg bd and placebo bd. Week 8 and 22: assessment of ischemic-reperfusion injury with Technetium Annexin A5 Scintigraphy. Ischemic intervention: 10 minutes ischemia of the non-dominant arm with at the same time rhythmic contractions of the forearm and hand muscles.

Main study parameters/endpoints: Annexin targeting in the thenar muscle after ischemic exercise. The primary analysis is the difference in annexin targeting following 8 weeks of treatment with rosiglitazone 4 mg bd or placebo.

ELIGIBILITY:
Inclusion Criteria:

* At least 3 features of the metabolic syndrome (AHA/NHLBI).
* Willing and able to provide a signed and dated written informed consent.
* Men or postmenopausal women aged between 20 and 70 years.

Exclusion Criteria:

* Fasting glucose > 7,0 mmol/L or the use of hypoglycaemic agents. If fasting plasma glucose is between 6.1 and 7,0 mmol/L, an oral 75 g glucose test will be performed to exclude diabetes mellitus.
* Exposure to a PPAR-g agonist during the last 4 months or a documented significant hypersensitivity to a PPAR-g agonist.
* Participant in another study.
* Angina or heart failure (NYHA I-IV).
* Clinically significant liver disease (3 times the upper normal limit of ALAT, ASAT, AF, γGT or LDH)
* Clinically significant anemia (male Hb < 6,9 mmol/L, female < 6,25 mmol/L)
* Creatinin clearance < 40 mL/min
* Alcohol or drug abuse.
* Any physical inability to perform the exercise protocol.
* Administration of any radio pharmacon for research purposes in the previous 5 years.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2007-04; Primary Completion 2008-07 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Annexin targeting in the thenar muscle after ischemic exercise. The primary analysis is the difference in annexin targeting following 8 weeks of treatment with rosiglitazone 4 mg bd or placebo.

SECONDARY OUTCOMES:
The effect of rosiglitazone as compared to placebo on the HOMA-index.
Changes in vital signs, body weight, clinical laboratory parameters and adverse events monitoring during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Gerard A Rongen, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center, department pharmacology-Toxicology; Alexander JM Rennings, MD, Principal Investigator — Radboud University Nijmegen Medical Center, department of pharmacology-Toxicology; Paul Smits, MD, PhD, Study Director — Radboud University Nijmegen Medical Center, head of department of Parmacology-Toxicology
Locations (1):
- Clinical research Center Nijmegen, Nijmegen, Netherlands

REFERENCES:
- [Background] Grundy SM, Benjamin IJ, Burke GL, Chait A, Eckel RH, Howard BV, Mitch W, Smith SC Jr, Sowers JR. Diabetes and cardiovascular disease: a statement for healthcare professionals from the American Heart Association. Circulation. 1999 Sep 7;100(10):1134-46. doi: 10.1161/01.cir.100.10.1134. No abstract available. PMID 10477542
- [Background] Aronson D, Rayfield EJ, Chesebro JH. Mechanisms determining course and outcome of diabetic patients who have had acute myocardial infarction. Ann Intern Med. 1997 Feb 15;126(4):296-306. doi: 10.7326/0003-4819-126-4-199702150-00006. PMID 9036802
- [Background] Yue TL, Bao W, Gu JL, Cui J, Tao L, Ma XL, Ohlstein EH, Jucker BM. Rosiglitazone treatment in Zucker diabetic Fatty rats is associated with ameliorated cardiac insulin resistance and protection from ischemia/reperfusion-induced myocardial injury. Diabetes. 2005 Feb;54(2):554-62. doi: 10.2337/diabetes.54.2.554. PMID 15677515
- [Background] Rongen GA, Oyen WJ, Ramakers BP, Riksen NP, Boerman OC, Steinmetz N, Smits P. Annexin A5 scintigraphy of forearm as a novel in vivo model of skeletal muscle preconditioning in humans. Circulation. 2005 Jan 18;111(2):173-8. doi: 10.1161/01.CIR.0000151612.02223.F2. Epub 2004 Dec 27. PMID 15623546